CLINICAL TRIAL: NCT06252077
Title: Effect of Very Low Ketogenic Diet on Energy Metabolism in Women With Obesity
Brief Title: Very Low Ketogenic Diet and Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Alessio Basolo, Researcher, PhD, MD, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EECR
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Energy Metabolism

STUDY DESIGN:
Intervention Model Description: body weight loss
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- very low ketogenic diet (Experimental): patients with overweight and obesity in treatment for weight loss
  Interventions: Dietary Supplement: very low ketogenic diet

INTERVENTIONS:
Dietary Supplement: very low ketogenic diet — 1 month of active phase of very low ketogenic diet

SUMMARY:
This study aimed at evaluating the effectiveness of the active phase of a very low-calorie ketogenic diet in females with obesity lasting 28 days on body weight, body composition and energy metabolism using a metabolic chamber.

DETAILED DESCRIPTION:
Patients were recruited at the Obesity and Lipodystrophy Center, University Hospital of Pisa. Enrolled subjects underwent active phase of very low-calorie ketogenic diet within the metabolic chamber from day 0 for a duration of 4 weeks (day 0-28). On days 0, 7, and 28, patients underwent a 24-hour measurement of energy metabolism using the metabolic chamber. On the day of exit from the chamber measurement of body composition was conducted using total-body densitometry (Lunar iDXA; GE Healthcare).

ELIGIBILITY:
Inclusion Criteria:

* overweight and obesity

Exclusion Criteria:

* Type 1 and type 2 diabetes mellitus
* endocrine disorders
* asthma or pulmonary conditions
* cardiovascular disease
* gastrointestinal disease
* liver disease
* kidney diseases
* anemia (hemoglobin < 11 g/dL)
* leucopenia (white blood cells < 4,000/mcL)
* thrombocytopenia (platelets < 150,000/mcL)
* central nervous system disorders
* neurodegenerative diseases
* psychiatric disorders
* eating disorders
* alcohol abuse and substance dependence
* pregnancy
* lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2025-03-16 (Actual)

PRIMARY OUTCOMES:
measure of energy expenditure | 1 month
  measures of energy expenditure (in kilocalories) will be assessed by using the metabolic chamber, 24-hour whole room indirect calorimeter. Thus, the measures will be expressed in Kilocalories over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ferruccio Santini, MD, Principal Investigator — University of Pisa
Locations (1):
- University Hospital of Pisa, Endocrinology Unit, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No